CLINICAL TRIAL: NCT06554860
Title: Scapular Blackburn Stabilization Versus Proprioceptive Neuromuscular Facilitation in Subacromial Impingement Syndrome
Brief Title: Scapular Blackburn Stabilization Versus PNF in Impingement Syndrome
Acronym: impingment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Esmat Fouad Ebrahem, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Blackburn versus PNF
Record Dates: First submitted 2024-07-18; First posted 2024-08-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Impingement Syndrome
Keywords: Scapular Blackburn stabilization; Scapular PNF
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental. (Experimental): receive a scapular PNF exercise program in addition to conventional Exercise ,
  Interventions: Other: scapular Blackburn stabilization plus exercise
- Experimental (Experimental): receive a scapular Blackburn stabilization exercises in addition to conventional Exercise
  Interventions: Other: PNF plus Exercise
- control group (Other): Exercise only
  Interventions: Other: exercise only

INTERVENTIONS:
Other: scapular Blackburn stabilization plus exercise — scapular Blackburn stabilization
  Arms: Experimental.
Other: PNF plus Exercise — PNF plus Exercise
  Arms: Experimental
Other: exercise only — Exercise only
  Arms: control group

SUMMARY:
purpose of study to Aim to investigate effect(s) of scapular Blackburn stabilization exercises compared toscapular proprioceptive neuromuscular facilitation (SPNF) exercise in addition to conventional exercises on shoulder pain, function, shoulder,sacpular ROM, scapular muscle strength and scapular orientation in patients with sub acromial impingement syndrome

Participants will be randomly allocated to three groups as follow:

Group A (n=17): will receive a program of conventional exercise include rotator cuff strengthening ,stretching for posterior capsule and stretching for pectoralis minor for 18 sessions (3 sessions per week for six weeks) Group B (n=17): will receive a scapular PNF exercise program in addition to conventional Exercise with the same frequency. Group C (n=17): will receive a scapular Blackburn stabilization exercises in addition to conventional Exercise with the same frequency

DETAILED DESCRIPTION:
Sub-acromial impingement syndrome(SIS) is the most frequent cause of pain and overhead reach limitation in the shoulder area. It occurs when there is impingement of tendons or bursa in the shoulder from bones of the shoulder. Intrinsic and extrinsic factors that contribute to the development of SIS include inflammation in the supra humeral space, inhibition of the rotator cuff muscles, degeneration of the rotator cuff tendons, abnormal scapular position and kinematics. Currently SIS covers a range of pathologies from sub acromial bursitis to rotator cuff tendinopathy and full thickness rotator cuff tears.

The trial will guide physical therapists in selecting effective therapeutic interventions for patients with SAIS and scapular dyskinesia, aiming to reduce the number of treatment sessions, speed up recovery, and improve shoulder pain and functional abilities.

Scapular Blackburn stabilization exercise minimizes excessive superior translation of the humeral head in the glenoid fossa during elevation and subacromial space impingement, consequently addressing shoulder impingement. It also strengthens the scapulothoracic and rotator cuff muscles and decreases muscle imbalance.

Proprioceptive Neuromuscular Facilitation has been described as a comprehensive rehabilitation concept, promoting motor learning, motor control, strength and mobility.

This comprehensive rehabilitation approach includes task-oriented training with manual facilitation aimed at motor learning and motor control.

therefore, what are the effects of scapular Blackburn stabilization and PNF techniques in addition to conventional exercises on shoulder pain, function, shoulder ROM, scapular muscle strength, and scapular orientation in patients with sub acromial impingement syndrome?

ELIGIBILITY:
Inclusion Criteria:

* 1. Fifty one Male and female patients with SIS and aged between 30-50.

  2. Body mass index (BMI) 18.5-29.9 kg/m2.

  3. patients complaining primary shoulder impingement.

  4. patients with altered scapular resting positions with scapular dyskinesia with positive lateral scapular slide test.

  5- patients will be included at least three special tests positive from the following tests:

A-Hawkins-Kennedy Impingement Test:

B-Neer"s Impingement Test:

C- "Empty Can" or Jobe Test D-painful arc test

E-External rotation resistance test

F-Cross-body adduction test

G-Drop arm sign

Exclusion Criteria:

* 1- Neurological deficit affecting the shoulder function during daily activities.

  2-Cervical disc pathology.

  3- Brain injures.

  4- Fractures in the upper limb

  5-Undergone shoulder surgery

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
shoulder pain and functional disability | Assessment procedure will be performed pre intervention and post third and sixth week of treatment
  Shoulder pain and disability index., minimum number 0=mean No pain and No disabilities and maximum number 10=mean highest pain and maximum disability
A-shoulder flexion ROM B- shoulder external rotation C-shoulder internal rotation | Assessment procedure will be performed pre intervention and post third and sixth week of treatment
  Digital Inclinometer.
selective muscle strength on: A- upper trapezius B- middle trapezius C-lower trapezius. D- serrates anterior | Assessment procedure will be performed pre intervention and post third and sixth week of treatment
  -Lafayette Hand-held dynamometer
scapula orientation | Assessment procedure will be performed pre intervention and post third and sixth week of treatment
  lateral scapular slide test

CONTACTS AND LOCATIONS:
Overall Officials: Enas F. Youssef, Prof.Dr, Principal Investigator — chair person of Department of Physical therapy for Musculoskeletal Disorder and its Surgery
Locations (1):
- faculty of physical therapy Cairo university, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Aceituno-Gomez J, Avendano-Coy J, Gomez-Soriano J, Garcia-Madero VM, Avila-Martin G, Serrano-Munoz D, Gonzalez-Gonzalez J, Criado-Alvarez JJ. Efficacy of high-intensity laser therapy in subacromial impingement syndrome: a three-month follow-up controlled clinical trial. Clin Rehabil. 2019 May;33(5):894-903. doi: 10.1177/0269215518824691. Epub 2019 Jan 23. PMID 30672303
- [Background] AlHarbi Y. Anatomical Variations in the Pectoralis Minor Muscle Origin and Insertion: A Systematic Review. Cureus. 2023 Oct 1;15(10):e46329. doi: 10.7759/cureus.46329. eCollection 2023 Oct. PMID 37916251
- [Background] Abdul-Karim S, Abdul-Hamid MS, Ho CA, Ling J. Validity, Reliability and Responsiveness of the Malay Shoulder Pain and Disability Index (M-SPADI) for Patients with Shoulder Pain. Malays Orthop J. 2023 Mar;17(1):160-171. doi: 10.5704/MOJ.2303.019. PMID 37064621
- [Background] Alsanawi HA, Alghadir A, Anwer S, Roach KE, Alawaji A. Cross-cultural adaptation and psychometric properties of an Arabic version of the Shoulder Pain and Disability Index. Int J Rehabil Res. 2015 Sep;38(3):270-5. doi: 10.1097/MRR.0000000000000118. PMID 25954858
- [Background] An DI, Park JE, Lee CH, Kim SY. Reliability of scapular upward rotation and anterior-posterior tilt measurements using a modified digital inclinometer in patients with subacromial impingement syndrome. J Back Musculoskelet Rehabil. 2021;34(5):837-843. doi: 10.3233/BMR-200080. PMID 33935062
- [Background] Breckenridge JD, McAuley JH. Shoulder Pain and Disability Index (SPADI). J Physiother. 2011;57(3):197. doi: 10.1016/S1836-9553(11)70045-5. PMID 21843839
- [Background] Bot SD, Terwee CB, van der Windt DA, Bouter LM, Dekker J, de Vet HC. Clinimetric evaluation of shoulder disability questionnaires: a systematic review of the literature. Ann Rheum Dis. 2004 Apr;63(4):335-41. doi: 10.1136/ard.2003.007724. PMID 15020324
- [Background] Boykin RE, Friedman DJ, Zimmer ZR, Oaklander AL, Higgins LD, Warner JJ. Suprascapular neuropathy in a shoulder referral practice. J Shoulder Elbow Surg. 2011 Sep;20(6):983-8. doi: 10.1016/j.jse.2010.10.039. Epub 2011 Feb 1. PMID 21277806
- [Background] Blennow K, Brody DL, Kochanek PM, Levin H, McKee A, Ribbers GM, Yaffe K, Zetterberg H. Traumatic brain injuries. Nat Rev Dis Primers. 2016 Nov 17;2:16084. doi: 10.1038/nrdp.2016.84. PMID 27853132
- [Background] Boettcher CE, Ginn KA, Cathers I. The 'empty can' and 'full can' tests do not selectively activate supraspinatus. J Sci Med Sport. 2009 Jul;12(4):435-9. doi: 10.1016/j.jsams.2008.09.005. Epub 2008 Dec 2. PMID 19054712
- [Background] Cools AM, Vanderstukken F, Vereecken F, Duprez M, Heyman K, Goethals N, Johansson F. Eccentric and isometric shoulder rotator cuff strength testing using a hand-held dynamometer: reference values for overhead athletes. Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3838-3847. doi: 10.1007/s00167-015-3755-9. Epub 2015 Aug 21. PMID 26294055
- [Background] Celik D, Dirican A, Baltaci G. Intrarater reliability of assessing strength of the shoulder and scapular muscles. J Sport Rehabil. 2012 Feb 29;21(1):1-5. doi: 10.1123/jsr.2012.TR3. Print 2012 Feb 1. PMID 22495260
- [Background] Cools AM, Cambier D, Witvrouw EE. Screening the athlete's shoulder for impingement symptoms: a clinical reasoning algorithm for early detection of shoulder pathology. Br J Sports Med. 2008 Aug;42(8):628-35. doi: 10.1136/bjsm.2008.048074. Epub 2008 Jun 3. PMID 18523035
- [Background] Consigliere P, Haddo O, Levy O, Sforza G. Subacromial impingement syndrome: management challenges. Orthop Res Rev. 2018 Oct 23;10:83-91. doi: 10.2147/ORR.S157864. eCollection 2018. PMID 30774463
- [Background] Curtis T, Roush JR. The Lateral Scapular Slide Test: A Reliability Study of Males with and without Shoulder Pathology. N Am J Sports Phys Ther. 2006 Aug;1(3):140-6. PMID 21522226
- [Background] Cools AM, Dewitte V, Lanszweert F, Notebaert D, Roets A, Soetens B, Cagnie B, Witvrouw EE. Rehabilitation of scapular muscle balance: which exercises to prescribe? Am J Sports Med. 2007 Oct;35(10):1744-51. doi: 10.1177/0363546507303560. Epub 2007 Jul 2. PMID 17606671
- [Background] Cools AM, Declercq G, Cagnie B, Cambier D, Witvrouw E. Internal impingement in the tennis player: rehabilitation guidelines. Br J Sports Med. 2008 Mar;42(3):165-71. doi: 10.1136/bjsm.2007.036830. Epub 2007 Dec 10. PMID 18070811
- [Background] Cibulka MT, Weissenborn D, Donham M, Rammacher H, Cuppy P, Ross SA. A new manual muscle test for assessing the entire trapezius muscle. Physiother Theory Pract. 2013 Apr;29(3):242-8. doi: 10.3109/09593985.2012.718856. Epub 2012 Sep 7. PMID 22957845
- [Background] Curtis L, Rea W, Smith-Willis P, Fenyves E, Pan Y. Adverse health effects of outdoor air pollutants. Environ Int. 2006 Aug;32(6):815-30. doi: 10.1016/j.envint.2006.03.012. Epub 2006 May 30. PMID 16730796
- [Background] Desai V, Stambulic T, Daneshvar P, Bicknell RT. Lower trapezius tendon transfer for irreparable rotator cuff injuries: a scoping review. JSES Rev Rep Tech. 2022 Sep 30;3(1):1-9. doi: 10.1016/j.xrrt.2022.08.006. eCollection 2023 Feb. PMID 37588064
- [Background] Dougherty J, Walmsley S, Osmotherly PG. Passive range of movement of the shoulder: a standardized method for measurement and assessment of intrarater reliability. J Manipulative Physiol Ther. 2015 Mar-Apr;38(3):218-24. doi: 10.1016/j.jmpt.2014.11.006. Epub 2015 Feb 20. PMID 25704219
- [Background] Day JM, Jones T, Eiben K, Berger Y. Scapular motion is accelerated in asymptomatic individuals with dyskinesis: An observational study. J Bodyw Mov Ther. 2021 Apr;26:134-140. doi: 10.1016/j.jbmt.2020.12.034. Epub 2021 Feb 6. PMID 33992234
- [Background] de Winter AF, Heemskerk MA, Terwee CB, Jans MP, Deville W, van Schaardenburg DJ, Scholten RJ, Bouter LM. Inter-observer reproducibility of measurements of range of motion in patients with shoulder pain using a digital inclinometer. BMC Musculoskelet Disord. 2004 Jun 14;5:18. doi: 10.1186/1471-2474-5-18. PMID 15196309
- [Background] Ellenbecker TS, Cools A. Rehabilitation of shoulder impingement syndrome and rotator cuff injuries: an evidence-based review. Br J Sports Med. 2010 Apr;44(5):319-27. doi: 10.1136/bjsm.2009.058875. PMID 20371557
- [Background] Edouard P, Degache F, Oullion R, Plessis JY, Gleizes-Cervera S, Calmels P. Shoulder strength imbalances as injury risk in handball. Int J Sports Med. 2013 Jul;34(7):654-60. doi: 10.1055/s-0032-1312587. Epub 2013 Feb 26. PMID 23444085
- [Background] Escamilla RF, Hooks TR, Wilk KE. Optimal management of shoulder impingement syndrome. Open Access J Sports Med. 2014 Feb 28;5:13-24. doi: 10.2147/OAJSM.S36646. eCollection 2014. PMID 24648778
- [Background] Greving K, Dorrestijn O, Winters JC, Groenhof F, van der Meer K, Stevens M, Diercks RL. Incidence, prevalence, and consultation rates of shoulder complaints in general practice. Scand J Rheumatol. 2012 Mar;41(2):150-5. doi: 10.3109/03009742.2011.605390. Epub 2011 Sep 21. PMID 21936616
- [Background] Ginn KA, Cohen ML. Exercise therapy for shoulder pain aimed at restoring neuromuscular control: a randomized comparative clinical trial. J Rehabil Med. 2005 Mar;37(2):115-22. doi: 10.1080/16501970410023443. PMID 15788347
- [Background] Ganderton C, Kinsella R, Watson L, Pizzari T. Getting more from standard rotator cuff strengthening exercises. Shoulder Elbow. 2020 Jun;12(3):203-211. doi: 10.1177/1758573219888829. Epub 2019 Dec 4. PMID 32565922
- [Background] Longo UG, Risi Ambrogioni L, Berton A, Candela V, Massaroni C, Carnevale A, Stelitano G, Schena E, Nazarian A, DeAngelis J, Denaro V. Scapular Dyskinesis: From Basic Science to Ultimate Treatment. Int J Environ Res Public Health. 2020 Apr 24;17(8):2974. doi: 10.3390/ijerph17082974. PMID 32344746
- [Background] Hughes P. The Neer sign and Hawkins-Kennedy test for shoulder impingement. J Physiother. 2011;57(4):260. doi: 10.1016/S1836-9553(11)70061-3. No abstract available. PMID 22093129
- [Background] Hopkins C, Fu SC, Chua E, Hu X, Rolf C, Mattila VM, Qin L, Yung PS, Chan KM. Critical review on the socio-economic impact of tendinopathy. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2016 Apr 22;4:9-20. doi: 10.1016/j.asmart.2016.01.002. eCollection 2016 Apr. PMID 29264258
- [Background] Harrington SE, Hoffman J, Katsavelis D. Measurement of Pectoralis Minor Muscle Length in Women Diagnosed With Breast Cancer: Reliability, Validity, and Clinical Application. Phys Ther. 2020 Mar 10;100(3):429-437. doi: 10.1093/ptj/pzz174. PMID 32043149
- [Background] Huang HY, Lin JJ, Guo YL, Wang WT, Chen YJ. EMG biofeedback effectiveness to alter muscle activity pattern and scapular kinematics in subjects with and without shoulder impingement. J Electromyogr Kinesiol. 2013 Feb;23(1):267-74. doi: 10.1016/j.jelekin.2012.09.007. Epub 2012 Nov 2. PMID 23123099
- [Background] Hwang M, Lee S, Lim C. Effects of the Proprioceptive Neuromuscular Facilitation Technique on Scapula Function in Office Workers with Scapula Dyskinesis. Medicina (Kaunas). 2021 Apr 1;57(4):332. doi: 10.3390/medicina57040332. PMID 33915824
- [Background] Hodgins JL, Rubenstein W, Kovacevic D, Padaki A, Jobin CM, Ahmad CS. Pectoralis Minor Contracture in Throwing Shoulders of Asymptomatic Adolescent Baseball Players. Orthop J Sports Med. 2017 Sep 20;5(9):2325967117728041. doi: 10.1177/2325967117728041. eCollection 2017 Sep. PMID 28975133
- [Background] Hoffman JR, Ratamess NA, Tranchina CP, Rashti SL, Kang J, Faigenbaum AD. Effect of protein-supplement timing on strength, power, and body-composition changes in resistance-trained men. Int J Sport Nutr Exerc Metab. 2009 Apr;19(2):172-85. doi: 10.1123/ijsnem.19.2.172. PMID 19478342
- [Background] Hussey JM, Nguyen QC, Whitsel EA, Richardson LJ, Halpern CT, Gordon-Larsen P, Tabor JW, Entzel PP, Harris KM. The reliability of in-home measures of height and weight in large cohort studies: Evidence from Add Health. Demogr Res. 2015 Jan-Jun;32:1081-1098. doi: 10.4054/DemRes.2015.32.39. PMID 26146486
- [Background] Hotta GH, Gomes de Assis Couto A, Cools AM, McQuade KJ, Siriani de Oliveira A. Effects of adding scapular stabilization exercises to a periscapular strengthening exercise program in patients with subacromial pain syndrome: A randomized controlled trial. Musculoskelet Sci Pract. 2020 Oct;49:102171. doi: 10.1016/j.msksp.2020.102171. Epub 2020 Jun 29. PMID 32861372
- [Background] Ishigaki T, Yoshino K, Hirokawa M, Sugawara M, Yamanaka M. Supraspinatus tendon thickness and subacromial impingement characteristics in younger and older adults. BMC Musculoskelet Disord. 2022 Mar 11;23(1):234. doi: 10.1186/s12891-022-05179-y. PMID 35277147
- [Background] Inui H, Osawa S, Mimori K. Coracoid process transfer and distal clavicle resection for chronic acromioclavicular separation. JSES Int. 2022 Oct 17;7(1):93-97. doi: 10.1016/j.jseint.2022.09.012. eCollection 2023 Jan. PMID 36820424
- [Background] IJspeert J, Kerstens HCJW, Janssen RMJ, Geurts ACH, van Alfen N, Groothuis JT. Validity and reliability of serratus anterior hand held dynamometry. BMC Musculoskelet Disord. 2019 Aug 7;20(1):360. doi: 10.1186/s12891-019-2741-7. PMID 31391035
- [Background] Kibler WB, Ludewig PM, McClure PW, Michener LA, Bak K, Sciascia AD. Clinical implications of scapular dyskinesis in shoulder injury: the 2013 consensus statement from the 'Scapular Summit'. Br J Sports Med. 2013 Sep;47(14):877-85. doi: 10.1136/bjsports-2013-092425. Epub 2013 Apr 11. PMID 23580420
- [Background] Kim MK, Lee JC, Yoo KT. The effects of shoulder stabilization exercises and pectoralis minor stretching on balance and maximal shoulder muscle strength of healthy young adults with round shoulder posture. J Phys Ther Sci. 2018 Mar;30(3):373-380. doi: 10.1589/jpts.30.373. Epub 2018 Mar 2. PMID 29581654
- [Background] Murphy RJ, Carr AJ. Shoulder pain. BMJ Clin Evid. 2010 Jul 22;2010:1107. PMID 21418673
- [Background] Karas V, Cole BJ, Wang VM. Role of biomechanics in rotator cuff pathology: North American perspective. Med Sport Sci. 2012;57:18-26. doi: 10.1159/000328871. Epub 2011 Oct 4. PMID 21986042
- [Background] Kevern MA, Beecher M, Rao S. Reliability of measurement of glenohumeral internal rotation, external rotation, and total arc of motion in 3 test positions. J Athl Train. 2014 Sep-Oct;49(5):640-6. doi: 10.4085/1062-6050-49.3.31. Epub 2014 Sep 4. PMID 25188316
- [Background] Karnawat S, Harikesavan K, Venkatesan P. Effect of Functional Scapular Stabilization Training on Function and Pain in Frozen Shoulder Syndrome: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2023 Feb;46(2):86-97. doi: 10.1016/j.jmpt.2023.05.008. Epub 2023 Jul 15. PMID 37452810
- [Background] Lin P, Yang M, Huang D, Lin H, Wang J, Zhong C, Guan L. Effect of proprioceptive neuromuscular facilitation technique on the treatment of frozen shoulder: a pilot randomized controlled trial. BMC Musculoskelet Disord. 2022 Apr 20;23(1):367. doi: 10.1186/s12891-022-05327-4. PMID 35443651
- [Background] Lowry V, Lavigne P, Zidarov D, Matifat E, Cormier AA, Desmeules F. A Systematic Review of Clinical Practice Guidelines on the Diagnosis and Management of Various Shoulder Disorders. Arch Phys Med Rehabil. 2024 Feb;105(2):411-426. doi: 10.1016/j.apmr.2023.09.022. Epub 2023 Oct 11. PMID 37832814
- [Background] Iida N, Taniguchi K, Watanabe K, Miyamoto H, Taniguchi T, Teramoto A, Katayose M. Effective stretching positions for the posterior shoulder capsule as determined by shear wave elastography. J Shoulder Elbow Surg. 2021 May;30(5):1186-1195. doi: 10.1016/j.jse.2020.08.021. Epub 2020 Sep 9. PMID 32919046
- [Background] Lee JH, Park SJ, Na SS. The effect of proprioceptive neuromuscular facilitation therapy on pain and function. J Phys Ther Sci. 2013 Jun;25(6):713-6. doi: 10.1589/jpts.25.713. Epub 2013 Jul 23. PMID 24259836
- [Background] Longo UG, Risi Ambrogioni L, Candela V, Berton A, Lo Presti D, Denaro V. Scapular Kinematics and Patterns of Scapular Dyskinesis in Rotator Cuff Tears: A Prospective Cohort Study. J Clin Med. 2023 Jun 4;12(11):3841. doi: 10.3390/jcm12113841. PMID 37298036
- [Background] Michener LA, Sharma S, Cools AM, Timmons MK. Relative scapular muscle activity ratios are altered in subacromial pain syndrome. J Shoulder Elbow Surg. 2016 Nov;25(11):1861-1867. doi: 10.1016/j.jse.2016.04.010. Epub 2016 Jun 30. PMID 27374236
- [Background] McQuade KJ, Borstad J, de Oliveira AS. Critical and Theoretical Perspective on Scapular Stabilization: What Does It Really Mean, and Are We on the Right Track? Phys Ther. 2016 Aug;96(8):1162-9. doi: 10.2522/ptj.20140230. Epub 2016 Feb 4. PMID 26847012
- [Background] Michener LA, Walsworth MK, Doukas WC, Murphy KP. Reliability and diagnostic accuracy of 5 physical examination tests and combination of tests for subacromial impingement. Arch Phys Med Rehabil. 2009 Nov;90(11):1898-903. doi: 10.1016/j.apmr.2009.05.015. PMID 19887215
- [Background] Mannava S, Plate JF, Whitlock PW, Callahan MF, Seyler TM, Koman LA, Smith TL, Tuohy CJ. Evaluation of in vivo rotator cuff muscle function after acute and chronic detachment of the supraspinatus tendon: an experimental study in an animal model. J Bone Joint Surg Am. 2011 Sep 21;93(18):1702-11. doi: 10.2106/JBJS.J.00184. PMID 21938374
- [Background] Motwani R, Kaliappan A, Chandrupatla M. Variant pectoralis minor muscle: a case study with clinical relevance. Anat Cell Biol. 2022 Dec 31;55(4):406-413. doi: 10.5115/acb.22.076. Epub 2022 Oct 20. PMID 36263504
- [Background] Oliver GD, Wasserberger K, de Swart A, Friesen K, Downs J, Bordelon N. Effects of Hip Range of Motion and Isometric Strength on Energy Flow during Windmill Softball Pitching. J Athl Train. 2021 Jan 22. doi: 10.4085/145-20. Online ahead of print. PMID 33480995
- [Background] Peteraitis T, Smedes F. Scapula motor control training with Proprioceptive Neuromuscular Facilitation in chronic subacromial impingement syndrome: A case report. J Bodyw Mov Ther. 2020 Jul;24(3):165-171. doi: 10.1016/j.jbmt.2020.03.005. Epub 2020 Mar 15. PMID 32825984
- [Background] Park SE, Wang JS. Effect of joint mobilization using KEOMT and PNF on a patient with CLBP and a lumbar transitional vertebra: a case study. J Phys Ther Sci. 2015 May;27(5):1629-32. doi: 10.1589/jpts.27.1629. Epub 2015 May 26. PMID 26157278
- [Background] Penning LI, De Bie RA, Leffers P, Weijers RE, Walenkamp GH. Empty can and drop arm tests for cuff rupture : Improved specificity after subacromial injection. Acta Orthop Belg. 2016 Aug;82(2):166-173. PMID 27682276
- [Background] Petersen SM, Wyatt SN. Lower trapezius muscle strength in individuals with unilateral neck pain. J Orthop Sports Phys Ther. 2011 Apr;41(4):260-5. doi: 10.2519/jospt.2011.3503. Epub 2011 Feb 2. PMID 21289453
- [Background] Paul A, Lewis M, Shadforth MF, Croft PR, Van Der Windt DA, Hay EM. A comparison of four shoulder-specific questionnaires in primary care. Ann Rheum Dis. 2004 Oct;63(10):1293-9. doi: 10.1136/ard.2003.012088. PMID 15361390
- [Background] Paraskevopoulos E, Papandreou M, Gliatis J. Reliability of assessment methods for scapular dyskinesis in asymptomatic subjects: A systematic review. Acta Orthop Traumatol Turc. 2020 Sep;54(5):546-556. doi: 10.5152/j.aott.2020.19088. PMID 33155568
- [Background] Ravichandran H, Janakiraman B, Gelaw AY, Fisseha B, Sundaram S, Sharma HR. Effect of scapular stabilization exercise program in patients with subacromial impingement syndrome: a systematic review. J Exerc Rehabil. 2020 Jun 30;16(3):216-226. doi: 10.12965/jer.2040256.128. eCollection 2020 Jun. PMID 32724778
- [Background] Rosa DP, Borstad JD, Pogetti LS, Camargo PR. Effects of a stretching protocol for the pectoralis minor on muscle length, function, and scapular kinematics in individuals with and without shoulder pain. J Hand Ther. 2017 Jan-Mar;30(1):20-29. doi: 10.1016/j.jht.2016.06.006. Epub 2016 Oct 18. PMID 27769843
- [Background] Roy JS, MacDermid JC, Woodhouse LJ. Measuring shoulder function: a systematic review of four questionnaires. Arthritis Rheum. 2009 May 15;61(5):623-32. doi: 10.1002/art.24396. PMID 19405008
- [Background] Singh H, Thind A, Mohamed NS. Subacromial Impingement Syndrome: A Systematic Review of Existing Treatment Modalities to Newer Proprioceptive-Based Strategies. Cureus. 2022 Aug 25;14(8):e28405. doi: 10.7759/cureus.28405. eCollection 2022 Aug. PMID 36171841
- [Background] Shadmehr A, Sarafraz H, Heidari Blooki M, Jalaie SH, Morais N. Reliability, agreement, and diagnostic accuracy of the Modified Lateral Scapular Slide test. Man Ther. 2016 Aug;24:18-24. doi: 10.1016/j.math.2016.04.004. Epub 2016 Apr 19. PMID 27317502
- [Background] Shadmehr A, Bagheri H, Ansari NN, Sarafraz H. The reliability measurements of lateral scapular slide test at three different degrees of shoulder joint abduction. Br J Sports Med. 2010 Mar;44(4):289-93. doi: 10.1136/bjsm.2008.050872. Epub 2008 Sep 23. PMID 18812417
- [Background] Struyf F, Nijs J, Mollekens S, Jeurissen I, Truijen S, Mottram S, Meeusen R. Scapular-focused treatment in patients with shoulder impingement syndrome: a randomized clinical trial. Clin Rheumatol. 2013 Jan;32(1):73-85. doi: 10.1007/s10067-012-2093-2. Epub 2012 Oct 2. PMID 23053685
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Toprak U, Ustuner E, Ozer D, Uyanik S, Baltaci G, Sakizlioglu SS, Karademir MA, Atay AO. Palpation tests versus impingement tests in Neer stage I and II subacromial impingement syndrome. Knee Surg Sports Traumatol Arthrosc. 2013 Feb;21(2):424-9. doi: 10.1007/s00167-012-1969-7. Epub 2012 Mar 28. PMID 22453312
- [Background] Tozzo MC, Ansanello W, Martins J, Zatiti SCA, de Oliveira AS. Inclinometer Reliability for Shoulder Ranges of Motion in Individuals With Subacromial Impingement Syndrome. J Manipulative Physiol Ther. 2021 Mar;44(3):236-243. doi: 10.1016/j.jmpt.2020.12.001. Epub 2021 Apr 27. PMID 33926742
- [Background] Takeno K, Glaviano NR, Norte GE, Ingersoll CD. Therapeutic Interventions for Scapular Kinematics and Disability in Patients With Subacromial Impingement: A Systematic Review. J Athl Train. 2019 Mar;54(3):283-295. doi: 10.4085/1062-6050-309-17. Epub 2019 Mar 4. PMID 30829536
- [Background] Viriyatharakij N, Chinkulprasert C, Rakthim N, Patumrat J, Ketruang B. Change of pectoralis minor length, and acromial distance, during scapular retraction at 60 degrees shoulder elevation. J Bodyw Mov Ther. 2017 Jan;21(1):53-57. doi: 10.1016/j.jbmt.2016.04.015. Epub 2016 Apr 29. PMID 28167190
- [Background] Villafane JH, Valdes K, Anselmi F, Pirali C, Negrini S. The diagnostic accuracy of five tests for diagnosing partial-thickness tears of the supraspinatus tendon: A cohort study. J Hand Ther. 2015 Jul-Sep;28(3):247-51; quiz 252. doi: 10.1016/j.jht.2015.01.011. Epub 2015 Feb 19. PMID 26003014
- [Background] Yaari LS, Mullaney MJ, Fukunaga T, Thein R, McHugh MP, Nicholas SJ. ASSESSMENT OF HUMERAL TORSION BY PALPATION IN BASEBALL PITCHERS: A VALIDATION STUDY. Int J Sports Phys Ther. 2020 Dec;15(6):1073-1079. doi: 10.26603/ijspt20201073. PMID 33344024